CLINICAL TRIAL: NCT02168439
Title: Double Blinded Randomized Controlled Trial of Intranasal Dexmedetomidine Versus Intranasal Midazolam as Anxiolysis Prior to Pediatric Laceration Repair in the Emergency Department
Brief Title: Intranasal Dexmedetomidine vs Intranasal Midazolam as Anxiolysis Prior to Pediatric Laceration Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Clinical and Translational Science Institute (CTSI) (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Desiree Neville, MD, M.D., Pediatric Emergency Medicine Fellow Physician, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRO13120431; UL1TR000005 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Laceration; Anxiety
Keywords: Dexmedetomidine; Midazolam
MeSH Terms: conditions — Lacerations; Anxiety Disorders | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Intranasal Dexmedetomidine 2 micrograms/kilogram once
  Interventions: Drug: Dexmedetomidine
- Midazolam (Experimental): Intranasal Midazolam 0.4 milligram/kilogram
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Midazolam
  Other Names: Versed
  Arms: Midazolam

SUMMARY:
The objective of this research study is to show superiority of intranasal dexmedetomidine to intranasal midazolam as anxiolysis prior to pediatric laceration repairs.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center
* Laceration <5 cm in total length
* Require simple suture laceration repair

Exclusion Criteria:

* Allergies/intolerance/contraindication to the study drugs
* Lacerations requiring complex (multilayer) repair or total laceration length>5cm

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Neville, MD, Principal Investigator — Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: Intranasal Dexmedetomidine 2 micrograms/kilogram once
  Dexmedetomidine: 20 patients enrolled, 20 underwent analysis
- Midazolam: Intranasal Midazolam 0.4 milligram/kilogram
  Midazolam: 20 patients enrolled, 18 underwent analysis
Period: Overall Study
Arm/Group | Dexmedetomidine | Midazolam
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: 38 patients were analyzed in total.
Groups:
- Dexmedetomidine: Intranasal Dexmedetomidine 2 micrograms/kilogram once
  Dexmedetomidine: .
- Midazolam: Intranasal Midazolam 0.4 milligram/kilogram
  Midazolam: .
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Midazolam | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Full Range); unit: years] | 3.44 [1.6 to 5.4] | 3.15 [1.0 to 5.4] | 3.21 [1.0 to 5.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38
Laceration length [Mean (Standard Deviation); unit: centimeters] | 1.59 (.87) | 1.44 (.73) | 1.52 (.79)

OUTCOME MEASURES:

1. Primary Outcome: mYPAS Score as Completed by Researchers to Assess Anxiety
Description: Primary outcome was the mYPAS scores at the time of positioning for procedure.
  mYPAS stands for modified Yale Preoperative anxiety scale. The scale is from minimum 23.3- maximum 100. Higher scores indicate higher anxiety. By prior characterization, scores less than or equal to 30 are classified as not anxious.
Time Frame: Day 1
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Dexmedetomidine | Midazolam
Number analyzed (Participants) | 20 | 18
units on a scale | 23.3 [23.3 to 30.8] | 36.3 [32.5 to 38.8]

2. Secondary Outcome: mYPAS Scores at Other Time Points
Description: mYPAS stands for modified Yale Preoperative anxiety scale. The scale is from minimum 23.3- maximum 100. Higher scores indicate higher anxiety. By prior characterization, scores less than or equal to 30 are classified as not anxious.
Time Frame: Day 1
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Dexmedetomidine | Midazolam
Number analyzed (Participants) | 20 | 18
units on a scale
  Baseline Anxiety | 48.8 [36.7 to 82.5] | 47.1 [40.0 to 51.3]
  Anxiety at Wound Washout | 42.5 [23.3 to 88.3] | 47.1 [34.2 to 67.5]
  Anxiety at First Stitch Placement | 23.3 [23.3 to 89.2] | 35.4 [31.3 to 52.9]

3. Secondary Outcome: VAS for Anxiety as Completed by Caregiver and Observer
Description: VAS, Visual Analog Scale for anxiety. Scale from 0-10 written on a 10 cm horizontal line with the extremes labeled as no anxiety to very anxious.
  Vertical line is drawn on the scale at the level of anxiety. The distance was measured.
  Higher numbers equal higher anxiety.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Midazolam
Number analyzed (Participants) | 20 | 18
units on a scale
  VAS Baseline | 3.8 (2.9) | 3.5 (3.5)
  VAS Position | 1.7 (2.9) | 1.6 (2.4)
  VAS Recovery | .7 (1.6) | 1.2 (1.6)

4. Other Pre Specified Outcome: Procedure Completion
Description: note of whether the procedure was able to be completed
Time Frame: Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Dexmedetomidine | Midazolam
Number analyzed (Participants) | 20 | 18
percentage of participants | 100 | 100

5. Other Pre Specified Outcome: Need for Procedural Sedation
Description: Whether the patient required procedural sedation for completion of the procedure
Time Frame: Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Dexmedetomidine | Midazolam
Number analyzed (Participants) | 20 | 18
percentage of participants | 0 | 0

6. Other Pre Specified Outcome: Anxiolysis Satisfaction
Description: Likert scale parent, child life and proceduralist survey
  5 point likert scale asking how satisfied the parent or proceduralist is with the anxiolysis from the medication.
  1 being not satisfied at all, 3 neutral, 5 very satisfied.
Time Frame: Day 1
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Midazolam
Number analyzed (Participants) | 20 | 18
units on a scale
  Parent Satisfaction | 5 (1.3) | 5 (1.1)
  Proceduralist Satisfaction | 4.5 (1.3) | 5 (1.4)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Midazolam
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=20) | Midazolam (N=18)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — vomiting after going home from repair
fall (Nervous system disorders) | 0 (0) | 1 (1) — fall after repair while in the ED

LIMITATIONS AND CAVEATS:
2 patients not included in the midazolam group: one for equipment malfunction leading to no data collected and the second due to weight error resulting in the patient receiving over twice the dose. Both recognized around the time of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No